CLINICAL TRIAL: NCT02459496
Title: Dietary Strategies to Improve Metabolism and Body Weight in Type 2 Diabetes
Brief Title: Diabetes Nutrition Algorithms in Patients With Overt Diabetes Mellitus
Acronym: DiNA-D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: German Center for Diabetes Research (Other); California Walnut Company (Other); Institute for Cereal Processing GmbH/Institut für Getreideverarbeitung (IGV) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Director of the Department for Clinical Nutrition, German Institute of Human Nutrition
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DiNA-D
Record Dates: First submitted 2015-03-23; First posted 2015-06-02 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes; NAFLD; Obesity; Dyslipoproteinaemia; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Obesity; Dyslipidemias; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low-carb diet, followed by conventional DGE diet (Active Comparator): subjects receive dietary consulting for a first phase of 3 weeks, being represented by a very-low calory low-carb ketogenic diet (VLCKD, below 40 g carbs per day), followed by an isocaloric or moderate hypocaloric low-carb diet (below 40 kcal% carbs per day)
  Interventions: Behavioral: dietary consulting and advise
- very-low calory diet, followed by conventional diet (Active Comparator): subjects receive dietary consulting for a first phase of 3 weeks, being represented by a very-low calory diet (VLCD; MODIFAST substitute, approx. 1200 kcal/day), followed by a conventional isocaloric or moderate hypocaloric diet under DGE guidelines
  Interventions: Behavioral: dietary consulting and advise

INTERVENTIONS:
Behavioral: dietary consulting and advise — first phase: 3 weeks of very-low calory diet (low-carb or normo-carb) second phase: 49 weeks of eucaloric diet under DGE guidelines

SUMMARY:
Basic treatment of type 2 diabetes should focus on diet, physical activity and lifestyle. Nevertheless, in early and late stage of T2DM, lifestyle intervention is mostly substituted by pharmacological intervention, although lifestyle modification and dietary treatment would be favourable.

The researchers therefore investigate dietary strategies such as low-carb and very-low calory diets regarding their potential to improve metabolism and body weight in (mostly) long-term T2DM patients.

DETAILED DESCRIPTION:
Basic treatment of type 2 diabetes should focus on diet, physical activity and lifestyle. Nevertheless, in early and late stage of T2DM, lifestyle intervention is mostly substituted by pharmacological intervention, although lifestyle modification and dietary treatment would be favourable.

The researchers therefore investigate dietary strategies such as low-carb diets and very-low calory diets regarding their potential to improve metabolism and body weight in (mostly) long-term T2DM patients.

An intensive intervention of 3 weeks is followed by an 11-month maintenance phase to consolidate metabolic improvements.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects
* 18-79 years old
* type 2 diabetes

Exclusion Criteria:

* renal insufficiency
* anaemia
* immunosuppression
* previous symptomatic cancer diagnosis
* acute cardiovascular disease (stroke, coronary syndrome)
* pregnancy and lactation
* severe psychiatric disorders
* corticoid or other immunosuppressive therapy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
change in insulin secretion (glucagon stimulation test) | 3 weeks, 1 year
  change in insulin secretion (glucagon stimulation test)
change in hepatic fat content (MR-S) | 3 weeks, 1 year
  change in hepatic fat content (MR-S)
change in insulin secretion in the mixed-meal tolerance test (MMTT) - combined parameter | 3 weeks, 1 year
  change in insulin secretion in the mixed-meal tolerance test (MMTT) - combined parameter
change in insulin sensitivity in the mixed-meal tolerance test (MMTT) - combined parameter | 3 weeks, 1 year
  change in insulin sensitivity in the mixed-meal tolerance test (MMTT) - combined parameter
change in blood glucose profile in the mixed-meal tolerance test (MMTT) - combined parameter | 3 weeks, 1 year
  change in blood glucose profile in the mixed-meal tolerance test (MMTT) - combined parameter

SECONDARY OUTCOMES:
inflammatory reaction in subcutaneous adipose tissue (SCAT analysis on protein and RNA level - IL-1; IL1beta, IL-6) | 3 weeks, 1 year
  inflammatory reaction in subcutaneous adipose tissue (SCAT analysis on protein and RNA level)
change in parameters of peripheral - vibration threshold, thermal sensitivity and pain thresholds | 3 weeks, 1 year
  peripheral neuropathy
change in parameters of autonomic neuropathy - measures of cardio-autonomic neuropathy (SANN, MSDD) | 3 weeks, 1 year
  autonomic neuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Andreas F.H. Pfeiffer, Prof. Dr. med., Principal Investigator — German Institute of Human Nutrition
Locations (2):
- Germany (2):
  - German Institut for Human Nutrition; Department for Clinical Nutrition, Bergholz-Rehbrücke, Brandenburg
  - German Institute for Human Nutrition, Department for Clinical Nutrition, Berlin